CLINICAL TRIAL: NCT00007995
Title: Phase 2 Study Of High Dose Chemotherapy Followed By Autologous Hematopoietic Stem Cell Support In Patients With Multiple Myeloma And Primary Light Chain Amyloidosis
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplant in Treating Patients Who Have Multiple Myeloma or Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068361; CPMC-IRB-7328; CPMC-CAMP-009; NCI-G00-1882
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2007-07

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Interferon-alpha; sargramostim; Busulfan; Cyclophosphamide; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Biological: sargramostim
Drug: busulfan
Drug: cyclophosphamide
Drug: melphalan
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well chemotherapy and peripheral stem cell transplant work in treating patients with multiple myeloma or primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with multiple myeloma or primary systemic amyloidosis treated with high-dose chemotherapy with autologous hematopoietic stem cell support.
* Determine the toxicity of this regimen in these patients.
* Determine the disease-free survival and overall survival of patients with multiple myeloma treated with this regimen.

OUTLINE: Patients are stratified according to disease response to prior treatment (responsive vs refractory or relapsed) and diagnosis (multiple myeloma vs primary systemic amyloidosis).

Following a course of induction chemotherapy, patients receive filgrastim (G-CSF) subcutaneously (SC) daily until the completion of peripheral blood stem cell (PBSC) harvesting. Patient who do not mobilize sufficient cells undergo bone marrow harvest.

Patients receive melphalan IV over 30 minutes on days -2 and -1. Half of the stored PBSCs and/or bone marrow is reinfused on day 0. Patients receive sargramostim (GM-CSF) daily beginning on day 0 and continuing until blood counts recover. Patients with primary systemic amyloidosis who are not responding to or are unable to tolerate treatment do not proceed to the second course of therapy.

Within 4-6 weeks after receiving melphalan, patients receive oral busulfan on days -8 to -5 followed by cyclophosphamide IV continuously on days -4 and -3. The remaining half of PBSCs and/or bone marrow is reinfused on day 0. Patients receive GM-CSF daily beginning on day 0 and continuing until blood counts recover.

Within 4-12 weeks after receiving the second course of high-dose chemotherapy, multiple myeloma patients receive maintenance therapy consisting of interferon alfa SC 3 days a week, after blood counts recover.

Patients are followed every 3 months for 1 year and then annually for 5 years.

PROJECTED ACCRUAL: Approximately 60-75 patients (25 for responsive disease stratum, 25 for refractory or relapsed disease stratum, and 10-25 for primary systemic amyloidosis stratum) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma OR
* Primary systemic amyloidosis resulting in significant organ dysfunction and decreased quality of life
* Complete or partial response after standard chemotherapy
* Primary refractory or relapsed multiple myeloma after first-line treatment with standard chemotherapy
* Ineligible for higher priority national or institutional clinical studies

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2 times normal

Renal:

* Creatinine less than 2.5 mg/dL or on stable hemodialysis

Cardiovascular:

* LVEF at least 45%

Pulmonary:

* DLCO at least 60% of predicted OR
* Approval by pulmonologist

Other:

* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Concurrent participation in gene therapy trials allowed

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent steroids as antiemetics during chemotherapy
* No concurrent anticancer hormonal therapy

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent barbiturates or acetaminophen during chemotherapy
* Concurrent participation in supportive care trials allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 1999-07; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Disease-free survival at 2 years (patients with responsive disease)

SECONDARY OUTCOMES:
Duration of hematologic toxicity
Time to an absolute neutrophil count
Platelet independence

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Hesdorffer, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York, United States